CLINICAL TRIAL: NCT05306314
Title: A Study to Understand the Treatment Patterns in Patients With Chronic Bacterial Prostatitis (Category II), Chronic Pelvic Pain (Category IIIA, IIIB)Treataprost Added to Standard Antibiotic Treatment in Real-life Clinical Practice
Brief Title: Retrospective Chart Review of Treataprost Added to Antibiotic Treatment in Patients With Chronic Prostatitis
Acronym: Treataprost
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: GMG Grand Medical (Other)
Collaborators: Gama CRO Tıbbi İlaç Araştırma Org.Tic.Ltd.Şti (Unknown)
Responsible Party: Sponsor
Other Study IDs: GMG.22.TRT.01
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-02

CONDITIONS: Quality of Life; Infection, Bacterial; PSA; Prostatitis
MeSH Terms: conditions — Bacterial Infections; Prostatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TREATAPROST 0 mL( BID- 10mL*2) PO: Treataprost 10 mL ( 5 mL 2*1- PO ) 42 days Generic Name : Treatarost Advance Dosage Form: Suspension, vials of 250 mL Dosage : 250 mL Frequency : 2*1 (BID) Duration: 42 days (6 weeks) Administration:Oral administration before meals 30 minutes as 20 mL(10mL*2)
  Interventions: Dietary Supplement: TREATAPROST
- Antibiotic Treatment (1*1) PO + NSAID (PRN) PO ya da SUPP: Levolon 500 mg ( 1*1 -PO) 28 daANTIBIOTIC TREATMENT Levolon 500 mg ( 1*1 - PO) 28 days (4 weeks) Dosage Form:Film-coated tablet Dosage : 500 mg Frequency : 1*1 Duration: 28 days (4 weeks) Administration:It should be taken orally, without chewing, with a sufficient amount of water. The tablets can be taken during or between meals.
  NSAID Diclomec 75 mg ( PRN- PO )- 28 days (4 weeks) Dosage Form:Tablet Dosage : 75 mg Frequency : PRN Duration: 28 days (4 weeks as per needed) Administration:It should be taken orally, without chewing, with a sufficient amount of water. The tablets can be taken during or between meals.
  Interventions: Dietary Supplement: TREATAPROST

INTERVENTIONS:
Dietary Supplement: TREATAPROST — oral administration before meals 30 minutes
  Other Names: Treatarost Advance

SUMMARY:
Multicenter, Retrospectivecohort study in patients with Chronic Prostatitis, Chronic Bacterial Prostatitis (Category II) and Chronic Pelvic Pain Syndrome (Category IIIA, IIIB) and 140 patients without other significant comorbidities will be participated.

The aim of the study is to collect post-treatment data to evaluate inflammation, infection status and quality of life with standard antibiotic therapy with NSAID and added Treataprost effect.

DETAILED DESCRIPTION:
This study will be conducted in Patients with Confirmed Chronic Prostatitis and the datas of these patients will be recorded.

In real clinical practice, the data of patients who received Treataprost in addition to antibiotic therapy with NSAIDs will be recorded.

This is a non-invasive retrospective cohort study.

The primary endpoint of this study is:

* To determine the socio-demographic (age, educational status, lifestyle) characteristics of cases with Chronic Prostatitis, Chronic Bacterial Prostatitis (Category II) and Chronic Pelvic Pain Syndrome (Category IIIA, IIIB)
* Treataprost added to standard antibiotic therapy and NSAID in clinical practice, Chronic Prostatitis, Chronic in patients with Bacterial Prostatitis (Category II) and Chronic Pelvic Pain Syndrome (Category IIIA, IIIB) understanding treatment patterns

The secondary endpoint of this study is:

* The aim of the study will to evaluated gather detailed information about the effect on quality of life of Treataprost given with standard antibiotic therapy and NSAID.
* It will be collected gather detailed information the infection status after post treatment Treataprost given with standard antibiotic therapy and NSAID

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years old and male.
* The participant must be willing and competent to give written informed consent. If the subject is unable to consent on his behalf, a legally acceptable representative (ie, acceptable to the International Council for Harmonization [ICH] and local law as appropriate) must give informed consent on his behalf.
* Chronic Prostatitis, Chronic Bacterial Prostatitis (Category II) and Chronic Pelvic Pain Syndrome (Category IIIA, IIIB) diagnosed with standard antibiotic therapy with NSAID and antibiotic therapy with NSAID together with Treataprost patients

Exclusion Criteria:

* In patients with Chronic Prostatitis, Chronic Bacterial Prostatitis (Category II) and Chronic Pelvic Pain Syndrome (Category IIIA, IIIB) not receiving any treatment
* For Chronic Prostatitis, Chronic Bacterial Prostatitis (Category II) and Chronic Pelvic Pain Syndrome (Category IIIA, IIIB) taking an herbal preparation other than Treataprost in addition to standard antibiotic therapy and NSAID
* Patients who have participated in any clinical trial and received an investigational product
* Patients who did not give written informed consent

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-probability samples
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
To determine the socio-demographic (age, educational status, lifestyle) characteristics of cases with Chronic Prostatitis, Chronic Bacterial Prostatitis (Category II) and Chronic Pelvic Pain Syndrome (Category IIIA, IIIB) | once
  Determining the relationship between the disease and collecting socio-demographic information such as age, education level, lifestyle
Treataprost added to standard antibiotic therapy and NSAID in clinical practice, Chronic Prostatitis, Chronic in patients with Bacterial Prostatitis (Category II) and Chronic Pelvic Pain Syndrome (Category IIIA, IIIB) understanding treatment patterns | once
  Collecting data on Treataprost treatment added to standard antibiotic treatment and NSAID in clinical practice

SECONDARY OUTCOMES:
The aim of the study will to evaluated gather detailed information about the effect on quality of life of Treataprost given with standard antibiotic therapy and NSAID. | Once
  To collect gather detailed information qualirt of life after post treatment
• It will be collected gather detailed information the infection status after post treatment Treataprost given with standard antibiotic therapy and NSAID | once
  To collect gather detailed information the infection status after post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Coşkun Kaya, Ass.Prof.Dr., Principal Investigator — TR Ministry of Health Eskişehir City Hospital; Gökhan Temeltaş, Prof.Dr., Principal Investigator — Manisa Celal Bayar University Hafsa Sultan Hospital; Cabir Alan, Prof. Dr., Principal Investigator — Çanakkale Onsekiz Mart University; Taylan Oksay, Prof.Dr., Principal Investigator — Süleyman Demirel University Faculty of Medicine
Locations (4):
- Turkey (Türkiye) (4):
  - 18 Mart University Faculty of Medicines, Çanakkale
  - TR Ministry of Health Eskişehir City Hospital, Eskişehir
  - Süleyman Demirel University Faculty of Medicines, Isparta
  - Manisa Celal Bayar University Hafsa Sultan Hospital, Manisa

IPD SHARING:
Plan to Share IPD: Undecided
IPD plan is not clear as the decision has not been performed yet. The IPD plan will be entered.

REFERENCES:
- [Result] Erdemir F, Parlaktaş BS, Uluocak N. "Prostatitlerin Patofizyolojisi, Tanısı, Tedavisi ve Değerlendirilmesindeki Yenilikler. Üroloji Bülteni. 2007;18(4):147-155.
- [Result] von Staden H. Herophilus, Herophilus Chalcedonius, The art of medicine in early Alexandria: Edition, Translation and Essays. Cambridge: Cambridge University Press, 1989.
- [Result] Stutzman RE, Walsh PC. In: Suprapubic and retropubik prostatectomy, 6th ed. Walsh PC, Retik AB, Stamey TA, Vaughan ED Jr, editors. Philadelphia: WB Saunders Co.; 1992. p.2851-6.
- [Result] Clemens JQ, Stephens-Shields AJ, Newcomb C, Rodriguez LV, Lai HH, Bradley CS, Naliboff BD, Griffith JW, Taple BJ, Gupta P, Afari N, Harte SE, Strachan E, Guo W, Landis JR. Correlates of 1-Year Change in Quality of Life in Patients with Urologic Chronic Pelvic Pain Syndrome: Findings from the Multidisciplinary Approach to the Study of Chronic Pelvic Pain (MAPP) Research Network. J Urol. 2020 Oct;204(4):754-759. doi: 10.1097/JU.0000000000001080. Epub 2020 Apr 15. PMID 32294397
- [Result] Clemens JQ, Meenan RT, O'Keeffe Rosetti MC, Kimes T, Calhoun EA. Prevalence of and risk factors for prostatitis: population based assessment using physician assigned diagnoses. J Urol. 2007 Oct;178(4 Pt 1):1333-7. doi: 10.1016/j.juro.2007.05.140. Epub 2007 Aug 16. PMID 17706722
- [Result] McNaughton Collins M, Pontari MA, O'Leary MP, Calhoun EA, Santanna J, Landis JR, Kusek JW, Litwin MS; Chronic Prostatitis Collaborative Research Network. Quality of life is impaired in men with chronic prostatitis: the Chronic Prostatitis Collaborative Research Network. J Gen Intern Med. 2001 Oct;16(10):656-62. doi: 10.1111/j.1525-1497.2001.01223.x. PMID 11679032
- [Result] Krieger JN, Nyberg L Jr, Nickel JC. NIH consensus definition and classification of prostatitis. JAMA. 1999 Jul 21;282(3):236-7. doi: 10.1001/jama.282.3.236. No abstract available. PMID 10422990
- [Result] Schaeffer AJ, Wendel EF, Dunn JK, Grayhack JT. Prevalence and significance of prostatic inflammation. J Urol. 1981 Feb;125(2):215-9. doi: 10.1016/s0022-5347(17)54976-9. No abstract available. PMID 7206060
- [Result] Khan FU, Ihsan AU, Khan HU, Jana R, Wazir J, Khongorzul P, Waqar M, Zhou X. Comprehensive overview of prostatitis. Biomed Pharmacother. 2017 Oct;94:1064-1076. doi: 10.1016/j.biopha.2017.08.016. Epub 2017 Aug 16. PMID 28813783
- [Result] Calhoun EA, McNaughton Collins M, Pontari MA, O'Leary M, Leiby BE, Landis JR, Kusek JW, Litwin MS; Chronic Prostatitis Collaborative Research Network. The economic impact of chronic prostatitis. Arch Intern Med. 2004 Jun 14;164(11):1231-6. doi: 10.1001/archinte.164.11.1231. PMID 15197050
- [Result] Krieger JN, Riley DE, Cheah PY, Liong ML, Yuen KH. Epidemiology of prostatitis: new evidence for a world-wide problem. World J Urol. 2003 Jun;21(2):70-4. doi: 10.1007/s00345-003-0329-0. Epub 2003 Apr 24. PMID 12712363
- [Result] Nickel JC, Downey JA, Nickel KR, Clark JM. Prostatitis-like symptoms: one year later. BJU Int. 2002 Nov;90(7):678-81. doi: 10.1046/j.1464-410x.2002.03007.x. PMID 12410746
- [Result] Habermacher GM, Chason JT, Schaeffer AJ. Prostatitis/chronic pelvic pain syndrome. Annu Rev Med. 2006;57:195-206. doi: 10.1146/annurev.med.57.011205.135654. PMID 16409145
- [Result] Nickel JC, Downey J, Hunter D, Clark J. Prevalence of prostatitis-like symptoms in a population based study using the National Institutes of Health chronic prostatitis symptom index. J Urol. 2001 Mar;165(3):842-5. PMID 11176483
- [Result] Coker TJ, Dierfeldt DM. Acute Bacterial Prostatitis: Diagnosis and Management. Am Fam Physician. 2016 Jan 15;93(2):114-20. PMID 26926407
- [Result] Workshop Committee of the National Institute of Diabetes and Digestive and Kidney Disease (NIDDK). Chronic Prostatitis workshop 1995: Bethesda, Maryland.
- [Result] Nickel JC, Teichman JM, Gregoire M, Clark J, Downey J. Prevalence, diagnosis, characterization, and treatment of prostatitis, interstitial cystitis, and epididymitis in outpatient urological practice: the Canadian PIE Study. Urology. 2005 Nov;66(5):935-40. doi: 10.1016/j.urology.2005.05.007. PMID 16286098
- [Result] Kobayashi I, Ikawa K, Nakamura K, Nishikawa G, Kajikawa K, Yoshizawa T, Watanabe M, Kato Y, Zennami K, Kanao K, Tobiume M, Yamada Y, Mitsui K, Narushima M, Morikawa N, Sumitomo M. Penetration of piperacillin-tazobactam into human prostate tissue and dosing considerations for prostatitis based on site-specific pharmacokinetics and pharmacodynamics. J Infect Chemother. 2015 Aug;21(8):575-80. doi: 10.1016/j.jiac.2015.04.015. Epub 2015 May 14. PMID 26050020
- [Result] Nickel JC. Prostatitis: evolving management strategies. Urol Clin North Am. 1999 Nov;26(4):737-51. doi: 10.1016/s0094-0143(05)70215-9. PMID 10584615
- [Result] Gratzke C, Bachmann A, Descazeaud A, Drake MJ, Madersbacher S, Mamoulakis C, Oelke M, Tikkinen KAO, Gravas S. EAU Guidelines on the Assessment of Non-neurogenic Male Lower Urinary Tract Symptoms including Benign Prostatic Obstruction. Eur Urol. 2015 Jun;67(6):1099-1109. doi: 10.1016/j.eururo.2014.12.038. Epub 2015 Jan 19. PMID 25613154
- [Result] McVary KT, Roehrborn CG, Avins AL, Barry MJ, Bruskewitz RC, Donnell RF, Foster HE Jr, Gonzalez CM, Kaplan SA, Penson DF, Ulchaker JC, Wei JT. Update on AUA guideline on the management of benign prostatic hyperplasia. J Urol. 2011 May;185(5):1793-803. doi: 10.1016/j.juro.2011.01.074. Epub 2011 Mar 21. PMID 21420124
- [Result] de la Rosette JJ, Hubregtse MR, Karthaus HF, Debruyne FM. Results of a questionnaire among Dutch urologists and general practitioners concerning diagnostics and treatment of patients with prostatitis syndromes. Eur Urol. 1992;22(1):14-9. doi: 10.1159/000474715. PMID 1425844
- [Result] Yang J, Liu L, Xie HW, Ginsberg DA. Chinese urologists' practice patterns of diagnosing and treating chronic prostatitis: a questionnaire survey. Urology. 2008 Sep;72(3):548-51. doi: 10.1016/j.urology.2008.03.061. Epub 2008 Jul 2. PMID 18597833
- [Result] Moon TD. Questionnaire survey of urologists and primary care physicians' diagnostic and treatment practices for prostatitis. Urology. 1997 Oct;50(4):543-7. doi: 10.1016/S0090-4295(97)00308-7. PMID 9338729
- [Result] Schaeffer AJ, Landis JR, Knauss JS, Propert KJ, Alexander RB, Litwin MS, Nickel JC, O'Leary MP, Nadler RB, Pontari MA, Shoskes DA, Zeitlin SI, Fowler JE Jr, Mazurick CA, Kishel L, Kusek JW, Nyberg LM; Chronic Prostatitis Collaborative Research Network Group. Demographic and clinical characteristics of men with chronic prostatitis: the national institutes of health chronic prostatitis cohort study. J Urol. 2002 Aug;168(2):593-8. PMID 12131316
- [Result] Pontari MA, Joyce GF, Wise M, McNaughton-Collins M; Urologic Diseases in America Project. Prostatitis. J Urol. 2007 Jun;177(6):2050-7. doi: 10.1016/j.juro.2007.01.128. PMID 17509285
- [Result] Hans R. Larsen, William R. Ware, The Prostate and Its Problems, published by: International Health News
- [Result] Shoskes DA, Thomas KD, Gomez E. Anti-nanobacterial therapy for men with chronic prostatitis/chronic pelvic pain syndrome and prostatic stones: preliminary experience. J Urol. 2005 Feb;173(2):474-7. doi: 10.1097/01.ju.0000150062.60633.b2. PMID 15643213
- [Result] Shoskes DA, Zeitlin SI, Shahed A, Rajfer J. Quercetin in men with category III chronic prostatitis: a preliminary prospective, double-blind, placebo-controlled trial. Urology. 1999 Dec;54(6):960-3. doi: 10.1016/s0090-4295(99)00358-1. PMID 10604689
- [Result] Celep Ali M. Kronik Pelvik Ağrı Sendromlu Hastaların Psikiyatrik Hastalıklar Açısından Değerlendirilmesi. Uzmanlık Tezi , Tokat: Gazi Osman Paşa Ünİ. Tıp Fakültesi, Aile Hekimliği ABD, 2007
- [Result] Steenkamp V, Gouws MC, Gulumian M, Elgorashi EE, van Staden J. Studies on antibacterial, anti-inflammatory and antioxidant activity of herbal remedies used in the treatment of benign prostatic hyperplasia and prostatitis. J Ethnopharmacol. 2006 Jan 3;103(1):71-5. doi: 10.1016/j.jep.2005.07.007. Epub 2005 Aug 24. PMID 16122891
- [Result] Paulis G. Inflammatory mechanisms and oxidative stress in prostatitis: the possible role of antioxidant therapy. Res Rep Urol. 2018 Sep 17;10:75-87. doi: 10.2147/RRU.S170400. eCollection 2018. PMID 30271757
- [Result] Stolarczyk M, Piwowarski JP, Granica S, Stefanska J, Naruszewicz M, Kiss AK. Extracts from Epilobium sp. herbs, their components and gut microbiota metabolites of Epilobium ellagitannins, urolithins, inhibit hormone-dependent prostate cancer cells-(LNCaP) proliferation and PSA secretion. Phytother Res. 2013 Dec;27(12):1842-8. doi: 10.1002/ptr.4941. Epub 2013 Feb 25. PMID 23436427
- [Result] Yoshida T, Yoshimura M, Amakura Y. Chemical and Biological Significance of Oenothein B and Related Ellagitannin Oligomers with Macrocyclic Structure. Molecules. 2018 Mar 2;23(3):552. doi: 10.3390/molecules23030552. PMID 29498647
- [Result] Kiss A, Kowalski J, Melzig MF. Effect of Epilobium angustifolium L. extracts and polyphenols on cell proliferation and neutral endopeptidase activity in selected cell lines. Pharmazie. 2006 Jan;61(1):66-9. PMID 16454210
- [Result] Tolmacheva AA, Rogozhin EA, Deryabin DG. Antibacterial and quorum sensing regulatory activities of some traditional Eastern-European medicinal plants. Acta Pharm. 2014 Jun;64(2):173-86. doi: 10.2478/acph-2014-0019. PMID 24914718
- [Result] Todd A. Linsenmeyer MD et al, Non-Antibiotic Alternatives for the Treatment of Urinary Tract Infections Following Spinal Cord Injury, Manuscript for Journal of Spinal Cord Medicine, 2005, Source of funding: The New Jersey Commission on Spinal Cord Research (NJCSCR)
- [Result] Christiansen BA, Bhatti S, Goudarzi R, Emami S. Management of Osteoarthritis with Avocado/Soybean Unsaponifiables. Cartilage. 2015 Jan;6(1):30-44. doi: 10.1177/1947603514554992. PMID 25621100
- [Result] Lequesne M, Maheu E, Cadet C, Dreiser RL. Structural effect of avocado/soybean unsaponifiables on joint space loss in osteoarthritis of the hip. Arthritis Rheum. 2002 Feb;47(1):50-8. doi: 10.1002/art1.10239. PMID 11932878
- [Result] Lamaud E, Robert AM, Wepierre J. Biochemical effects of unsaponifiable lipidic components of avocado and soya bean administered percutaneously on the connective tissue components of hairless rat skin. Int J Cosmet Sci. 1979 Aug;1(4):213-9. doi: 10.1111/j.1467-2494.1979.tb00216.x. PMID 19467069
- [Result] Heinecke LF, Grzanna MW, Au AY, Mochal CA, Rashmir-Raven A, Frondoza CG. Inhibition of cyclooxygenase-2 expression and prostaglandin E2 production in chondrocytes by avocado soybean unsaponifiables and epigallocatechin gallate. Osteoarthritis Cartilage. 2010 Feb;18(2):220-7. doi: 10.1016/j.joca.2009.08.015. Epub 2009 Sep 6. PMID 19748608
- [Result] de Oliveira GJ, de Paula LG, Spin-Neto R, Stavropoulos A, Spolidorio LC, Marcantonio E Jr, Marcantonio RA. Effect of avocado/soybean unsaponifiables on osseointegration: a proof-of-principle preclinical in vivo study. Int J Oral Maxillofac Implants. 2014 Jul-Aug;29(4):949-57. doi: 10.11607/jomi.3498. PMID 25032777
- [Result] Kishimoto H, Akagi M, Zushi S, Teramura T, Onodera Y, Sawamura T, Hamanishi C. Induction of hypertrophic chondrocyte-like phenotypes by oxidized LDL in cultured bovine articular chondrocytes through increase in oxidative stress. Osteoarthritis Cartilage. 2010 Oct;18(10):1284-90. doi: 10.1016/j.joca.2010.05.021. Epub 2010 Jul 13. PMID 20633688
- [Result] Hartmann RW, Mark M, Soldati F. Inhibition of 5 alpha-reductase and aromatase by PHL-00801 (Prostatonin(R)), a combination of PY102 (Pygeum africanum) and UR102 (Urtica dioica) extracts. Phytomedicine. 1996 Sep;3(2):121-8. doi: 10.1016/S0944-7113(96)80025-0. PMID 23194959
- [Result] Wagner H, Willer F, Samtleben R, Boos G. Search for the antiprostatic principle of stinging nettle (Urtica dioica) roots. Phytomedicine. 1994 Dec;1(3):213-24. doi: 10.1016/S0944-7113(11)80068-1. PMID 23195942
- [Result] Safarinejad MR. Urtica dioica for treatment of benign prostatic hyperplasia: a prospective, randomized, double-blind, placebo-controlled, crossover study. J Herb Pharmacother. 2005;5(4):1-11. PMID 16635963
- [Result] Klein-Bischoff U, Kaszkin-Bettag M, Heger PW, Sökeland J. Wirksamkeit des Brennnesselwurzel- Extraktes PU 240 bei BPH. Therapie Report aktuell, Uro-News 2007, 160(1-2): 1-6
- [Result] Rudick CN, Jiang M, Yaggie RE, Pavlov VI, Done J, Heckman CJ, Whitfield C, Schaeffer AJ, Klumpp DJ. O-antigen modulates infection-induced pain states. PLoS One. 2012;7(8):e41273. doi: 10.1371/journal.pone.0041273. Epub 2012 Aug 10. PMID 22899994
- [Result] Nickel JC, Downey J, Clark J, Casey RW, Pommerville PJ, Barkin J, Steinhoff G, Brock G, Patrick AB, Flax S, Goldfarb B, Palmer BW, Zadra J. Levofloxacin for chronic prostatitis/chronic pelvic pain syndrome in men: a randomized placebo-controlled multicenter trial. Urology. 2003 Oct;62(4):614-7. doi: 10.1016/s0090-4295(03)00583-1. PMID 14550427
- [Result] Zhou Z, Hong L, Shen X, Rao X, Jin X, Lu G, Li L, Xiong E, Li W, Zhang J, Chen Z, Pan J, Song B. Detection of nanobacteria infection in type III prostatitis. Urology. 2008 Jun;71(6):1091-5. doi: 10.1016/j.urology.2008.02.041. PMID 18538692
- [Result] Terai A, Ishitoya S, Mitsumori K, Ogawa O. Molecular epidemiological evidence for ascending urethral infection in acute bacterial prostatitis. J Urol. 2000 Dec;164(6):1945-7. PMID 11061888